CLINICAL TRIAL: NCT02677285
Title: Bioimpedance Based Monitoring of Operation Wound and Skin Graft Healing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other); Åbo Akademi University (Other); Turku PET Centre (Unknown); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R150095
Record Dates: First submitted 2016-01-25; First posted 2016-02-09 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Skin Graft; Closed Operation Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Skin graft: The bioimpedance measurement is done with a purpose built patch that has electrodes in contact with the wound and reference electrodes.
  Interventions: Other: Different type of wound
- Operation wound: The bioimpedance measurement is done with commercial electrodes places in healthy skin surrounding the wound.
  Interventions: Other: Different type of wound

INTERVENTIONS:
Other: Different type of wound

SUMMARY:
This study consists of two clinical series. With the first series investigators monitor the healing of skin grafts with bioimpedance measurements. The bioimpedance measurement is done with a purpose built patch that has electrodes in contact with the wound and reference electrodes.

In the second series the investigators monitor closed operational wounds (breast reconstruction surgery patients) with bioimpedance measurements. This series is also conducted with bioimpedance measurements but the wounds are operational wounds.

Both groups will have 20 patients.

DETAILED DESCRIPTION:
Objectives of the study:

1. The investigators will study how bioimpedance measurement results correlate with conventional wound healing monitoring.
2. The investigators will seek the best methods for handling, interpreting and presenting bioimpedance measurement results.
3. The investigators will find out if impedance measurement is applicable to clinical use.

ELIGIBILITY:
Inclusion Criteria:

* patients that have a skin graft operation made as part of their treatment
* patients that have breast reconstruction surgery made as part of their treatment

Exclusion Criteria:

* pregnancy
* patients with limited capacity to understand the information regarding the study
* patients with chronic skin disease on operation area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Plastic surgery and KEI2 wards at Tampere University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance data | 2 months
  Bioimpedance values between selected measuring points with different frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Kaartinen, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No